CLINICAL TRIAL: NCT07072247
Title: An Exploratory Clinical Study on the Safety and Efficacy of RN1201 Injection in the Treatment of Antibody-Mediated Diseases
Brief Title: RN1201 Injection in the Treatment of Antibody-Mediated Diseases
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Collaborators: Allorunning Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RN1201-Ab
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Refractory Immune-mediated Platelet Transfusion Refractoriness; Relapsed or Refractory Immune Thrombocytopenia
MeSH Terms: conditions — Recurrence; Purpura, Thrombocytopenic, Idiopathic | interventions — Antigens, CD19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allogeneic CAR-T cell therapy (Experimental): Antibody-Mediated Diseases treated with RN1201 Injection
  Interventions: Genetic: CD19 and BCMA-targeted allogeneic CAR-T cells

INTERVENTIONS:
Genetic: CD19 and BCMA-targeted allogeneic CAR-T cells — Lymphodepletion chemotherapy followed by CD19 and BCMA-targeted allogeneic CAR-T cells infusion
  Other Names: RN1201

SUMMARY:
This single-arm, open-label exploratory trial aims to evaluate the safety, feasibility, and preliminary efficacy of RN1201 Injection in patients with antibody-mediated diseases, including refractory immune-mediated platelet transfusion refractoriness (PTR) and relapsed or refractory immune thrombocytopenia (ITP). Patients will receive RN1201 cells infusion following lymphodepletion. The study will assess safety, response rates, B-cell depletion, and immune reconstitution. Exploratory analyses will examine in vivo persistence and activity of RN1201.

ELIGIBILITY:
Inclusion Criteria:

Inclusion: - specific for Refractory immune-mediated PTR:

1. Aged 16-65 years
2. Diagnosed with refractory immune-mediated PTR
3. Resistant to at least 3 standard therapies
4. Able to understand the study and consent
5. Projected survival time exceeding three months
6. Left Ventricular Ejection Fraction (LVEF) ≥0.5 (as measured by echocardiogram)
7. Creatinine <1.6 mg/dL
8. Aspartate Aminotransferase (AST) < three times the upper limit of normal
9. Total bilirubin <2.0 mg/dL
10. Karnofsky Performance Status (KPS) score ≥60.

Inclusion: -specific for Relapsed or Refractory Immune Thrombocytopenia

1. Written informed consent obtained;
2. Male or female patients aged 18 years or older on the day of informed consent signing;
3. Left Ventricular Ejection Fraction (LVEF) ≥50% with no pericardial effusion;
4. As assessed by the investigator, systemic treatment drugs (excluding supportive and symptomatic treatment, and prednisone at a daily dose of ≤10 mg or equivalent) can be discontinued prior to lymphodepletion preconditioning.
5. Historically diagnosed with primary immune thrombocytopenia (ITP) (based on the 2019 International Working Group for ITP and the American Society of Hematology (ASH));
6. At least two consecutive blood routine examinations showing reduced platelet count, with no significant abnormalities in blood cell morphology on peripheral blood smear microscopy;
7. At the screening visit, the subject has no splenomegaly;
8. Bone marrow examination: the bone marrow cytology of ITP patients is characterized by increased or normal megakaryocytes with maturation disorders (investigators may assess whether to accept previous bone marrow examination reports, and if previous reports are used, they must be kept as copies in the study documents);
9. The subject is a refractory ITP patient who has not responded to first-line treatment drugs, second-line thrombopoiesis-stimulating agents, and rituximab therapy, or who has undergone ineffective splenectomy or postoperative recurrence, and after re-evaluation of the diagnosis, is still confirmed to have ITP;
10. Relapsed ITP is defined as a decrease in platelet count to below 30×10⁹/L after an initial response to treatment, or to less than twice the baseline level, or the reappearance of bleeding symptoms.
11. The subject has received at least four weeks of the most recent treatment (non-biological background therapy, antimalarial monotherapy, antimalarial combined with oral glucocorticoids (OCS) and/or immunosuppressants, or combined therapy with OCS and/or immunosuppressants).

Exclusion Criteria:

Exclusion: - specific for Refractory immune-mediated PTR:

1. Uncontrolled active infection
2. Active hepatitis B or C infection
3. Patient has HIV or syphilis infection
4. Patient is pregnant or breastfeeding
5. Patient has a history of allogeneic hematopoietic stem cell transplantation (allo-HSCT)
6. Conventional treatment for antibody-mediated disease is effective
7. According to the New York Heart Association (NYHA) classification, patients with Class III/IV cardiovascular dysfunction
8. Other contraindications that make participation in this study unsuitable.

Exclusion: - specific for Relapsed or Refractory Immune Thrombocytopenia

1. Patients with the following conditions at the screening visit: Neutrophil count <1×10⁹/L; serum creatinine >1.5× upper limit of normal (ULN); immunoglobulin G (IgG) <5 g/L.
2. Subjects with Class III or IV heart failure according to the NYHA classification (see Appendix I)
3. Subjects with a history of epilepsy or other central nervous system diseases
4. Patients with active viral, bacterial or other infections requiring systemic treatment at the screening visit (including active or latent tuberculosis (TB) or SARS-CoV-2), or with a history of clinically significant recurrent infections (e.g., Bacillus infection);
5. Herpes or varicella-zoster virus infection within 12 weeks prior to the screening visit (particularly shingles);
6. Patients positive for HCV or HBsAg are excluded. HBcAb-positive patients are eligible only if HBsAg (regardless of anti-HBs status) and HBV DNA are negative;
7. Known history of primary or secondary immunodeficiency, or positive test results for HIV (ELISA and Western blot) at the screening visit;
8. Live vaccine or attenuated live vaccine administration within 4 weeks prior to the baseline visit;
9. Breastfeeding or pregnancy at the screening visit or prior to medication administration (positive serum or urine - β-hCG pregnancy test);
10. Females of childbearing potential and males whose partners are of childbearing potential must use medically approved contraception or abstain from sexual intercourse during the study treatment period and for at least 6 months after its completion. Females of childbearing potential must have a negative serum HCG test within 7 days before study enrollment and must not be breastfeeding;
11. History of malignancy, except for cured non-melanoma skin cancer, carcinoma in situ (e.g., cervical, breast, bladder, or prostate cancer), and tumors in complete remission for at least 3 years without evidence of recurrence;
12. Any severe and/or unstable pre-existing medical, psychiatric condition, or other disease that the investigator considers may interfere with the patient's efficacy, safety, informed consent, or compliance with the trial protocol;
13. Known hypersensitivity, intolerance, or contraindication to RN1201 or any excipients in the study drugs (including Fludarabine, Cyclophosphamide, and Tocilizumab), or a history of severe allergic reactions;
14. Participation in other investigational studies within 30 days prior to enrollment or within five half-lives of the study drug, whichever is longer.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 9 (Estimated)
Dates: Start 2025-07-10 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of treatment-emergent adverse events (TEAEs) and dose-limiting toxicities (DLTs) | within 4 weeks after infusion
  To characterize the safety of RN1201 Cells for Antibody-mediated Diseases

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From infusion up to 12 months post-treatment.
  The responses will be assessed based on changes of platelet count and incidence of bleeding events, according to predefined response criteria
Pharmacokinetic (PK) of RN1201 | From infusion up to 12 months post-treatment.
  Levels of RN1201 CAR-positive T cells in the blood and/or bone marrow
Pharmacodynamic (PD)-B cell depletion | From infusion up to 12 months post-treatment.
  Levels of B cells (direct and indirect measures) in the blood and/or bone marrow

IPD SHARING:
Plan to Share IPD: No